CLINICAL TRIAL: NCT02093260
Title: Phase II b Study of Immunogenicity and Safety of Flubio Vaccine in Infants and Children
Brief Title: Immunogenocity and Safety of Flubio (Influenza HA) Vaccine in Infants and Children (Bridging Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Influenza 0213
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Flubio Vaccine (Influenza HA); Infants; Children; Safety; Immunogenicity
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): Vaccine
  Flubio (Influenza HA) vaccine
  2 doses for infants and children (6 months - 8 years old)
  1 doses for children (9-11 years old)
  The vaccine will be given intramuscularly
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Flubio (Influenza HA) Vaccine
  The vaccine will be given intramuscularly.
  Other Names: Flubio

SUMMARY:
To Asses the Immunogenicity and Safety of Flubio (Influenza HA) Vaccine in Infants and Children (Bridging Study)

DETAILED DESCRIPTION:
Too see percentage of subjects with HI titer >= 1:40, 28 days after two doses in infants and children (6 months-8 years old) and one dose in children 9-11 years old for each strain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Parents have been informed properly regarding the study and signed the informed consent form
* Parents will commit themselves to comply with the instructions of the investigator and the schedule of the trial

Exclusion Criteria:

* Subjects concomitantly enrolled or scheduled to be enrolled in another trial
* Evolving mild, moderate, or severe illness, especially infectious diseases or fever (axillary temperature >=37oC)
* Known history of allergy to egg and/or chicken protein or any other component of the vaccines
* Known history of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
* Subject who has received a treatment likely to alter the immune response in the previous 4 weeks (intravenous immunoglobulins, blood-derived products or long term corticotherapy (>2 weeks)).
* Any abnormality or chronic disease justified by investigator that might interfere assessment of the trial objectives.
* Subjects has been immunized with influenza vaccine within 1 year
* Subjects receives any vaccination within 1 months before and after immunization of Flubio.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 405 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To asses the immunogenicity of Flubio vaccine 28 days after 2 doses immunization in infants and children (6 months-8 years of age) and 1 dose immunization in children (9-11 years of age) | 2 months
  Percentage of subjects with anti HI titer >=1:40

SECONDARY OUTCOMES:
To describe the seroconversion after 2 doses of Flubio vaccine in infants and children (6 months-8 years old) | 2 months
  Percentage subjects with increasing antibody titer >=4 times
To describe seroconversion after 1 dose of Flubio vaccine in children (9-11 years old) | 1 months
  Percentage of subjects with transition of seronegative to seropositive
To asses the safety of Flubio vaccine | 1-2 months
  Local and Systemic Reaction following immunization

CONTACTS AND LOCATIONS:
Overall Officials: Bernie Endyarni, MD, Principal Investigator — Department of Child Health, School of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Jatinegara Primary Health Center, Jakarta, Jakarta Special Capital Region
  - Primary School of SDN 01 Kampung Melayu, Jakarta, Jakarta Special Capital Region

REFERENCES:
- [Derived] Soedjatmiko S, Medise BE, Gunardi H, Sekartini R, Satari HI, Hadinegoro SR, Bachtiar NS, Sari RM. Immunogenicity and safety of a Trivalent Influenza HA vaccine in Indonesian infants and children. Vaccine. 2018 Apr 12;36(16):2126-2132. doi: 10.1016/j.vaccine.2018.02.114. Epub 2018 Mar 16. PMID 29551225